CLINICAL TRIAL: NCT03673540
Title: Using Ecological Momentary Interventions to Increase Skill Acquisition and Utilization
Brief Title: Acquisition and Utilization of Skills Using Innovative Smartphone Application for Regular Eating
Acronym: ACQUIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1802006074; R34MH116021 (NIH)
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Bulimia Nervosa; Bulimia; Binge Eating; Purging; Eating Disorder
Keywords: Bulimia Nervosa; Eating Disorder; Binge Eating; Bulimia; Purging
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT with smartphone application (EMI on) (Experimental): CBT with CBT+ smartphone application (EMI on)
  Interventions: Behavioral: CBT+ application

INTERVENTIONS:
Behavioral: CBT+ application — Smartphone application that comprises electronic self-monitoring of food intake, eating disorder behaviors, and mood and ecological momentary interventions
  Other Names: CBT+

SUMMARY:
The study seeks to evaluate the acceptability, feasibility, target engagement, and validity of an innovative smartphone application with ecological momentary interventions to augment cognitive behavioral therapy for bulimia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for bulimia nervosa or sub-threshold bulimia nervosa with subjective binge episodes (objective binge episodes or subjective binge episodes AND compensatory behaviors at least 1 time per week on average for the past 3 months)
* BMI >17.5
* Have a smartphone device
* Willing and able to use smartphone device to track food intake multiple times per day for 16 weeks

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next year
* Currently experiencing severe psychopathology that would limit their ability to engage in study (e.g. suicidality, substance use disorder, psychotic disorder)
* Have previously received a full trial of CBT for bulimia nervosa
* History of bariatric surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 61 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Binge and purge frequency assessed by the Eating Disorder Examination | Change from baseline assessment (before beginning treatment) to post-treatment assessment (16 weeks after baseline assessment)
  Frequency (number of days and number of instances) of binge eating and compensatory behaviors over the past 28 days assessed by the Eating Disorder Examination

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Assessed at weekly treatment sessions throughout treatment duration (16 weeks)
  The Eating Disorder Examination Questionnaire measures eating pathology. The EDE-Q yields four subscale scores: Restraint, Eating Concern, Shape Concern, and Weight Concern. The possible score range for each subscale is 0 to 6. The total score may also be reported (determined by averaging the subscale scores); the score range for the total score is also 0 to 6. For subscale scores and total score, higher scores indicate more severe pathology. The restraint sub-scale of the EDE-Q will be used to assess utilization of skills related to reducing dietary restraint.
Difficulties in Emotion Regulation Scale (DERS) | Assessed at weekly treatment sessions throughout treatment duration (16 weeks)
  The Difficulties in Emotion Regulation Scale is a self-report measure of emotional dysregulation. The DERS yields 6 subscale scores (Awareness, Clarity, Goals, Impulse, Nonacceptance, and Strategies) and a total score. The possible score range for each subscale is 3 to 15. The total score is computed by summing all 6 subscales, so the possible score range is 18 to 90. For all subscales and the total score, higher scores indicate greater difficulty in emotion regulation. The DERS will be used to assess utilization of skills related to increasing adaptive responses to cues.
Technology Acceptance Model Scale (TAMS) | Assessed at weekly treatment sessions throughout treatment duration (16 weeks)
  The Technology Acceptance Model Scale measures usefulness and ease of use of a technological product. The TAMS yields two subscale scores (usefulness and ease of use). The possible score range for each subscale is 6 to 49. Higher scores indicate greater usefulness and ease of use. The TAMS will be used to assess the perceived usefulness and perceived ease-of-use of the smartphone application to evaluate acceptability.
Feedback Questionnaire (FQ) | Assessed at weekly treatment sessions throughout treatment duration (16 weeks)
  The feedback questionnaire asks qualitative questions about the application. The feedback questionnaire does not report either subscale scores or a total score. The FQ will be used to obtain qualitative acceptability ratings.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Stratton Hall, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Presseller EK, Wilkinson ML, Trainor C, Lampe EW, Juarascio AS. Self-regulation deficits moderate treatment outcomes in a clinical trial evaluating just-in-time adaptive interventions as an augmentation to cognitive-behavioral therapy for bulimia-spectrum eating disorders. Int J Eat Disord. 2022 May;55(5):709-716. doi: 10.1002/eat.23695. Epub 2022 Feb 24. PMID 35212017
- [Derived] Presseller EK, Lampe EW, Michael ML, Trainor C, Fan SC, Juarascio AS. Latent trajectories of symptom change during cognitive-behavior therapy predict post-treatment worsening of symptoms: a preliminary examination among outpatients with bulimia-spectrum eating disorders. Eat Weight Disord. 2022 Aug;27(6):2257-2264. doi: 10.1007/s40519-021-01348-5. Epub 2022 Jan 4. PMID 34981464
- [Derived] Parker MN, Wilkinson ML, Hunt RA, Ortiz A, Manasse SM, Juarascio AS. Eating expectancies and hedonic hunger among individuals with bulimia-spectrum eating disorders who plan binge-eating episodes. Int J Eat Disord. 2022 Jan;55(1):120-124. doi: 10.1002/eat.23628. Epub 2021 Oct 13. PMID 34643949
- See also: For more information, send an email to EDresearch@drexel.edu or call (215) 553-7130 — http://drexel.edu/coas/academics/departments-centers/well-center/research/current-research-projects/